CLINICAL TRIAL: NCT03842644
Title: Postoperative Skin Surface Tension Relaxing in Prevention of Facial Surgical Skin Scarring: a Single Center, Perspective, Randomly, Controlled Clinical Trial.
Brief Title: Postoperative Skin Surface Tension Relaxing in Prevention of Facial Surgical Skin Scarring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: XiaoXi Lin (Other)
Responsible Party: Sponsor-Investigator, XiaoXi Lin, Professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Organization: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SH9H-2018-T65-2
Record Dates: First submitted 2019-02-02; First posted 2019-02-15 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Scar
Keywords: Tension Reduction
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tension Reduction (Experimental): Tension reduction device for 3 months post surgery
  Interventions: Device: Tension reduction device
- Control (No Intervention): No tension reduction

INTERVENTIONS:
Device: Tension reduction device — Continue using this device for 3 months post surgery.
  Other Names: Zipline Surgical Skin Closure Device
  Arms: Tension Reduction

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of early postoperative skin surface reduction in improving scar formation after facial surgery.

DETAILED DESCRIPTION:
Primary measurement: the mean scar width calculated by standard photos with rulers.

Secondary measure: the probability of scar hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* The incision is not shorter than 3cm
* Skin type is III/IV

Exclusion Criteria:

* Any medical history of facial surgery, not included injection therapy, external medication or fat graft
* Unsuitable for device use due to anatomical location of incision, eg. lips, eyelids and ear
* Patients with a history of keloid or family history of keloid
* Patients with serious skin disorders, eg. serious psoriasis or dermatitis
* Patients with severe systemic or congenital disease which may affect the patient's safety in this study

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2019-02-16 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
Scar width | through study completion, an average of 1 year
  scar width is measure by standard photo with ruler

SECONDARY OUTCOMES:
Hypertrophic scar rate | through study completion, an average of 1 year
  The onset of hypertrophic scar will be documented in the time of follow-up. The red and stiffness scar which higher than the surrounding skin surface will be considered as hypertrophic scar.
Patient and observer scar assessment scale score | through study completion, an average of 1 year
  Subscale 1: observer scar assessment scale (score range 5-50), the score 50 is considered as the worse outcome.
  Subscale 2: patient scar assessment scale (score range 5-50), the score 50 is considered as the worse outcome.
Vancouver Scar Scale | through study completion, an average of 1 year
  total score range from 0 to 14, the score14 is considered as the worse outcome
Relative side effect | through study completion, an average of 1 year
  The relative side effect will be documented in each time of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Lin, Professor, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China